CLINICAL TRIAL: NCT03158246
Title: Generic Zoledronic Acid Versus Original Zoledronic Acid: A Multicenter, Randomized, Open, Paralled-controlled Clinical Postmenopausal Osteoporotic Women Efficacy and Safety Research.
Brief Title: Generic Zoledronic Acid Versus Original Zoledronic Acid in Postmenopausal Osteoporotic Women
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cttq (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cttq-POWER
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: zoledronic acid; Yigu; Aclasta; Osteoporosis; Postmenopausal; BMD; fracture; Biochemical markers
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis; Fractures, Bone | interventions — Zoledronic Acid; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yigu Group (Experimental): a single 15-minute infusion of Generic Zoledronic Acid (Yigu®) (5 mg/100ml)
  600mg/d calcium and 925IU/d vitamin D for oral daily, 12 months
  Interventions: Drug: Generic Zoledronic Acid; Dietary Supplement: calcium; Dietary Supplement: vitamin D
- Aclasta Group (Active Comparator): a single 15-minute infusion of Original Zoledronic Acid (Aclasta®) (5 mg/100ml)
  600mg/d calcium and 925IU/d vitamin D for oral daily, 12 months
  Interventions: Drug: Original Zoledronic Acid; Dietary Supplement: calcium; Dietary Supplement: vitamin D

INTERVENTIONS:
Drug: Generic Zoledronic Acid — Generic Zoledronic Acid (Yigu®) 5mg/100ml injection
  Other Names: Yigu
  Arms: Yigu Group
Drug: Original Zoledronic Acid — Original Zoledronic Acid (Aclasta®) 5mg/100ml injection
  Other Names: Aclasta
  Arms: Aclasta Group
Dietary Supplement: calcium — 600mg/d calcium for oral daily
Dietary Supplement: vitamin D — 925IU/d vitamin D for oral daily

SUMMARY:
This study compares the efficacy and safety of generic zoledronic acid (Yigu®) and original zoledronic acid (Aclasta®) in the treatment of postmenopausal osteoporotic women in China. Four hundred and sixty-six subjects will be randomised (1:1ratio) to either Yigu® 5mg IV or Aclasta® 5mg IV treatment arms.

DETAILED DESCRIPTION:
A single infusion of intravenous zoledronic acid decreases bone turnover and improves bone density at 12 months in postmenopausal women with osteoporosis, and it significantly reduced the risk of vertebral fractures additionally.

In this research, the efficacy and safety of generic zoledronic acid injection in the treatment of postmenopausal osteoporosis will be evaluated, using original drug as control drug. It will provide evidence for reasonable clinical administrations.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women between the ages of 46 and 80（cessation of menses for 12 months for any reason）
* Subjects with osteoporosis diagnosed according to the World Health Organization (WHO) criteria：they had a BMD T-score of -2.5 or less at the spine or femoral neck；or they had low bone mass，defined as BMD T-score less than -1.0 and more than -2.5 at the spine or femoral neck，with the history of fragility fracture(Fracture site included vertebra, hip,proximal humera, distal radius, distal ulna)
* Subjects signed informed consent voluntarily

Exclusion Criteria:

* Any non-primary osteoporosis skeletal disease
* Subjects with abnormal hepatic function and renal function（alanine transaminase(ALT) and aspartate transaminase(AST) are 2 times higher than the upper limits of normal(ULN);plasma creatinine concentration and blood urea nitrogen are more than 1.5 ULN or calculated creatinine clearance less than 60 ml/min）
* Subjects with serum calcium greater than 2.75 mmol/L (11.0 mg/dL) or less than 2.00 mmol/L (8.0 mg/dL)
* Subjects with severe heart disease, blood disease, mental diseases
* Subjects with cancer and other serious progressive disease
* Prior therapy with bisphosphonates within 12 months before trial entry, prior therapy with parathyroid hormone 1-34 or 1-84, estrogen, selective estrogen receptor modulators, strontium more than 2 weeks within 6 months, prior therapy with oral or intravenous glucocorticoid more than 3 months within 6 months
* Subject is hypersensitivity to experimental drugs, comparator drugs and their metabolites
* Subjects who participated in other drugs or medical devices clinical studies as subjects within 3 months before this study
* Subjects judged unfit for this study by investigators

Ages: 46 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-02 (Estimated)

PRIMARY OUTCOMES:
Change in BMD T-scores | 12 months
  BMD T-scores (spine, hip and femoral neck) are determined versus baseline at the visits time

SECONDARY OUTCOMES:
Change in BMD T-scores | 6 months
  BMD T-scores (spine, hip and femoral neck) are determined versus baseline at the visits time
Change in Biochemical markers of bone turnover | 14 days, 6 months and 12 months
  Biochemical markers of bone turnover are determined versus baseline at the visits time. Including β-CTX and P1NP
Fractures | 12 months
  incidence of fracture of all parts

CONTACTS AND LOCATIONS:
Overall Officials: Xia Weibo, Study Chair — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Du Y, Yu W, Gou H, Lei Y, Zhang T, Tang W, Chen M, Li H, Cheng Q. Change in body temperature, not acute-phase reaction, predict anti-Osteoporosis efficacy after the first administration of Zoledronic acid: a prospective observational cohort study. BMC Musculoskelet Disord. 2024 Sep 2;25(1):694. doi: 10.1186/s12891-024-07781-8. PMID 39223504